CLINICAL TRIAL: NCT02037334
Title: Biomechanics Based Prediction of Preterm Delivery
Acronym: Softcervix
Status: Completed | Type: Observational
Sponsor: David Scheiner (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, David Scheiner, Sponsor-Investigator, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: KEK-ZH 2013-0244; 2013-MD-0036 (Other: Swissmedic)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Preterm Delivery
Keywords: Preterm delivery; Diagnostics; Biomechanics
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnancy
  Interventions: Device: Pregnolia System

INTERVENTIONS:
Device: Pregnolia System — No intervention is done except for measuring the stiffness of the cervix in pregnant women

SUMMARY:
Quantitative information on the biomechanical properties of the ecto-cervix in mid-pregnancy will be compared between women with term vs. preterm delivery. We aim to demonstrate that biomechanical data (ASP and CCI) might complement morphological data (CL) to improve prediction of preterm delivery. It is expected that women with preterm delivery will show stronger weakening of cervical tissue. Aspiration (ASP) and cervical CCI (cervical consistency index) measurements are performed at mid-pregnancy: detection at this time point is useful for therapy and biomechanical modifications are already significant so to enable differentiation by biomechanical measurements (ASP and CCI).

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women presenting at their mid pregnancy consultation (18+0 - 22+0 weeks of pregnancy) are eligible
* Signed informed consent after being informed is a prerequisite for enrollment.

Exclusion Criteria:

* Communication problems
* Missing consent
* Age<18
* Active bleeding / Premature Rupture of Membranes (PROM)
* Active genital infection
* Known carrier of HIV or Hepatitis B or C
* Placenta praevia
* Müllerian anomalies
* known or suspected non-compliance, drug or alcohol abuse
* cerclage
* use of pessary

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women at our institutions between 18+0/7 and 22+0/7 weeks of pregnancy and postpartum
Sampling Method: Non-Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Difference in cervical stiffness in women with/without preterm delivery | Measurements between 18+0/7 and 22+0/7 weeks of pregnancy and postpartum
  The biomechanical measurements and morphological data obtained at mid-pregnancy are compared between women with/without preterm delivery and are expected to significantly differ. The diagnostic power for preterm delivery of aspiration, CCI and the other factors will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: David A Scheiner, MD, Principal Investigator — University of Zurich
Locations (13):
- University Hospital of Leuven, Leuven, Belgium
- Switzerland (12):
  - Kantonsspital Aarau, Frauenklinik, Aarau
  - Kantonsspital Baden, Frauenklinik, Baden
  - Universitätsspital Basel, Frauenklinik, Basel
  - Kantonsspital Frauenfeld, Frauenklinik, Frauenfeld
  - Hôpitaux universitaires de Genève (HUG), Geneva
  - Kantonsspital Luzern, Frauenklinik, Lucerne
  - Kantonsspital Münsterlingen, Münsterlingen
  - Kantonsspital St. Gallen, Klinik für Gynäkologie und Geburtshilfe, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Praxis Zollikon, Zollikon
  - University Hospital of Zurich, Dept. OB/Gyn, Zurich
  - Stadtspital Triemli, Frauenklinik, Zurich